CLINICAL TRIAL: NCT03093298
Title: Searching for Altered Gene Expression in the Endocrine Secretome Following Roux-en-Y Gastric Bypass Surgery
Brief Title: The Endocrine Secretome After Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Filip Krag Knop (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor-Investigator, Filip Krag Knop, MD, PhD, professor, University Hospital, Gentofte, Copenhagen
Organization: University Hospital, Gentofte, Copenhagen (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H-6-2014-047
Record Dates: First submitted 2017-03-12; First posted 2017-03-28 (Actual); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Obesity, Morbid; Type2 Diabetes
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Obesity (Experimental): Enteroscopies with biopsy retrieval and mixed meal tests with blood sampling
  Interventions: Other: Enteroscopy with biopsy sampling and mixed meal test

INTERVENTIONS:
Other: Enteroscopy with biopsy sampling and mixed meal test — Enteroscopies with biopsy retrieval and mixed meal tests with blood sampling before and after Roux-en-Y gastric bypass surgery

SUMMARY:
Examination of the molecular phenotype and composition of endocrine cells in the gastrointestinal tract correlated to analyses of blood for hormones/analytes before and after Roux-en-Y gastric bypass surgery in morbidly obese individuals both with and without type 2 diabetes

DETAILED DESCRIPTION:
Enteroscopy was conducted during sedation with Propofol®. The pre-surgical sampling included biopsies retrieved from the stomach and at the expected site of anastomosis. During RYGB surgery, a ~1 cm gut tissue sample was removed at the site of anastomosis. The post-surgical enteroscopy ~3 months after RYGB surgery included biopsies taken from the gastric pouch, the alimentary limb, the biliopancreatic limb and common channel. One sample from each location was immersion-fixated in formalin for subsequent histological analyses and one sample was placed in a tube with RNA-preserving media for mRNA expression analysis. Remaining samples were snap-frozen and stored at -80°C until further processing.

Enteroendocrine cells were identified and isolated from biopsies obtained at several sites in the small intestine by using immunohistochemistry and laser capture technology. Isolated individual enteroendocrine cells were extensively characterised by next generation sequencing (Illumina NGS).

The participants also went through four mixed meal tests with blood sampling performed: before an 8 % diet-induced weight loss was initiated and one week before/one week after/3 months after RYGB surgery. Blood was sampled at several specific time points.

The plasma, serum and urine collected from study participants before and after RYGB surgery will be analysed for biomarkers/analytes and correlated with clinical data (weight, BMI, waist/hip ratio, blood pressure) and molecular phenotype found in gut samples.

To study changes in gut bacteria (microbiota) composition stool samples were collected during the study and will be analysed for microbiota composition by means of bacterial DNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Obese subjects referred for assessment of eligibility for RYGB surgery
* Age ≥25 and ≤ 60 years
* Able to understand written patient information and obtained signed informed consent
* Type 2 diabetes patients treated with lifestyle, metformin and/or sulfonylurea will be allowed participation.

Exclusion Criteria:

* Diagnosis of diabetes mellitus type 1
* Individuals being categorized as subjects with type 2 diabetes according to ADA 2014 criteria AND currently being treated with DPPIV inhibitors, GLP-1 agonists, insulin and/or SGLT2 inhibitors.
* Co-morbidities that, in the discretion of the investigators, exclude study participation such as chronic obstructive pulmonary disease (COPD) stage III, significant cardiac arrhythmias etc.
* Previous gastrointestinal surgery (excluding cholecystectomy and appendectomy).
* Gastrointestinal conditions making the subject unsuitable to participate in the study such as ulcerative colitis, Crohn´s disease, clinically significant food allergies, candidiasis etc.
* Chronic systemic inflammatory diseases (e.g,. rheumatoid arthritis) and other conditions significantly affecting inflammation status or immunoregulation (severe allergies, status post transplantation etc.)
* Chronic, planned or likely-to-be-required parenteral or oral corticosteroid medication during the study period, or (parenteral or oral) corticosteroid medication <4 weeks prior to screening
* Chronic infectious diseases such as hepatitis, HIV etc.
* Anaemia with a haemoglobin value 6.2 mmol/L (<10 g/dL) for women and 7.4 mmol/L (< 12 g/dL) for men at time of screening
* Clinically significant liver or kidney function impairment, or other laboratory findings leading to the diagnosis of clinically relevant disorders (severe thyroid dysfunction etc)
* Planned elective surgery (other than bariatric surgery) during the study period with the exception of dermatosurgical, ENT (ear, nose, throat) or dental procedures not requiring general anaesthesia and/or perioperative antibiotic treatment
* Abuse of alcohol and/or drugs, or any other co-existing conditions that will make the subject unsuitable to participate in the study, as deemed by the investigators
* Pregnancy or desire to become pregnant during the study period

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2014-12-12 (Actual); Primary Completion 2016-12-13 (Actual); Study Completion 2016-12-13 (Actual)

PRIMARY OUTCOMES:
Altered gene expression in the endocrine secretome following Roux-en-Y gastric bypass surgery | Each participant went through six study days (two mixed meal tests and one enteroscopy procedure before and after Roux-en-Y gastric bypass surgery, respectively)

CONTACTS AND LOCATIONS:
Overall Officials: Filip Knop, MD, prof., Principal Investigator — Gentofte Hospital, University of Copenhagen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gilliam-Vigh H, Suppli MP, Heimburger SMN, Lund AB, Knop FK, Ellegaard AM. Cholesin mRNA Expression in Human Intestinal, Liver, and Adipose Tissues. Nutrients. 2025 Feb 8;17(4):619. doi: 10.3390/nu17040619. PMID 40004948
- [Derived] Jorsal T, Christensen MM, Mortensen B, Nygaard EB, Zhang C, Rigbolt K, Wandall E, Langholz E, Friis S, Worm D, Floyd A, Helgstrand F, Stoving RK, Aldries AR, Juhl CB, Ostergaard T, Rydborg T, Forman JL, Sorensen F, Schmidt T, Falkenhahn M, Musholt PB, Theis S, Larsen PJ, Rehfeld JF, Vrang N, Jelsing J, Vilsboll T, Knop FK. Gut Mucosal Gene Expression and Metabolic Changes After Roux-en-Y Gastric Bypass Surgery. Obesity (Silver Spring). 2020 Nov;28(11):2163-2174. doi: 10.1002/oby.22973. PMID 33150746
- [Derived] Jorsal T, Wewer Albrechtsen NJ, Christensen MM, Mortensen B, Wandall E, Langholz E, Friis S, Worm D, Orskov C, Stoving RK, Andries A, Juhl CB, Sorensen F, Forman JL, Falkenhahn M, Musholt PB, Theis S, Larsen PJ, Holst JJ, Vrang N, Jelsing J, Vilsboll T, Knop FK. Investigating Intestinal Glucagon After Roux-en-Y Gastric Bypass Surgery. J Clin Endocrinol Metab. 2019 Dec 1;104(12):6403-6416. doi: 10.1210/jc.2019-00062. PMID 31276156